CLINICAL TRIAL: NCT05890391
Title: Time-Restricted Eating (16/8) and Energy-Restricted Diet: Effects on Diet Quality, Body Composition and Biochemical Parameters in Healthy Overweight Females
Brief Title: The Effect of Time-Restricted Eating on Nutritional Status
Acronym: TRE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Özge Mengi Çelik, assistant professor, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 86/2019
Record Dates: First submitted 2023-05-08; First posted 2023-06-06 (Actual); Last update posted 2023-06-06 (Actual); Status verified 2023-05

CONDITIONS: Energy Expenditure; Anthropometric Measure; Blood Pressure; Biochemical Markers; Healthy Eating Index
Keywords: time-restricted eating; diet quality; body composition; biochemical parameters
MeSH Terms: conditions — Intermittent Fasting

STUDY DESIGN:
Intervention Model Description: The female individuals were randomly divided into the TRE or ERD groups in an unbiased manner using a computer-generated block randomisation list.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Time-Restricted Eating (Experimental): Individuals in the TRE group applied a diet limited to 8 hours for 8 weeks.
  Interventions: Other: Time-Restricted Eating
- Energy-Restricted Diet (Experimental): Individuals in the ERD group followed a diet specially prepared for them for 8 weeks.
  Interventions: Other: Energy-Restricted Diet

INTERVENTIONS:
Other: Time-Restricted Eating — They were fed ad libitum between 10.00 a.m-06.00 p.m and fasted between 06.00 p.m-10.00 a.m.
  Arms: Time-Restricted Eating
Other: Energy-Restricted Diet — The total energy expenditure (TEE) of individuals was determined using the 'Resting Energy Expenditure (REE) x Physical Activity Level (PAL) ' formulation. 'TEE-500 kcal' formulation was used for the diet to be given to individuals.
  Arms: Energy-Restricted Diet

SUMMARY:
This study was planned to investigate the effect of TRE on the nutritional status and diet quality of individuals and to compare the effects of TRE and energy-restricted diet (ERD) in healthy overweight individuals. The female individuals were randomly divided into the TRE or ERD groups in an unbiased manner using a computer-generated block randomisation list. Individuals in the TRE group applied a diet limited to 8 hours for 8 weeks (16/8). They were fed ad libitum between 10.00 a.m-06.00 p.m and fasted between 06.00 p.m-10.00 a.m.No restrictions were imposed on the type and amount of food consumed during the feeding period. During the fasting period, individuals consumed water and non-energy drinks (tea, coffee, soda, etc.). Individuals in the ERD group followed a diet specially prepared for them for 8 weeks. At the first encounter with individuals, resting energy expenditure (REE) was measured by the indirect calorimetry method. Physical Activity Level (PAL) was determined by physical activity record. The total energy expenditure (TEE) of individuals was determined using the 'REE x PAL' formulation. 'TEE-500 kcal' formulation was used for the diet to be given to individuals. Individuals were not given a diet containing energy below the REE. Acceptable macronutrient distribution range (AMDR) were taken as dietary content. The diet given to individuals has 45-65% carbohydrate, 20-35% fat, 10-35% protein content. Nutritional habits of individuals were taken into consideration while planning the diet. Each individual consumed 3 main meals and the number of snacks was determined individually. Food exchange lists were given to individuals and nutrient changes were explained in detail. Anthropometric and body composition measurements of individuals were taken. The energy expenditure was measured using indirect calorimetry. Blood pressure and heart rate measurements were made. Biochemical parameters were evaluated and food consumption were taken. The quality of dietary intake was assessed using the Healthy Eating Index (HEI) -2015.

DETAILED DESCRIPTION:
The female individuals were randomly divided into the TRE or ERD groups in an unbiased manner using a computer-generated block randomisation list.

Individuals in the TRE group applied a diet limited to 8 hours for 8 weeks (16/8). They were fed ad libitum between 10.00 a.m-06.00 p.m and fasted between 06.00 p.m-10.00 a.m. No restrictions were imposed on the type and amount of food consumed during the feeding period.

Individuals in the ERD group followed a diet specially prepared for them for 8 weeks. At the first encounter with individuals, resting energy expenditure (REE) was measured by the indirect calorimetry method. Physical Activity Level (PAL) was determined by physical activity record. The total energy expenditure (TEE) of individuals was determined using the 'REE x PAL' formulation. 'TEE-500 kcal' formulation was used for the diet to be given to individuals. Individuals were not given a diet containing energy below the REE. Acceptable macronutrient distribution range (AMDR) were taken as dietary content. The diet given to individuals has 45-65% carbohydrate, 20-35% fat, 10-35% protein content. Nutritional habits of individuals were taken into consideration while planning the diet. Each individual consumed 3 main meals and the number of snacks was determined individually. Food exchange lists were given to individuals and nutrient changes were explained in detail.

Parameters to be evaluated at the beginning and end of the study

Anthropometric and body composition measurements The energy expenditure Blood pressure and heart rate measurements Biochemical parameters Food consumption The quality of dietary intake

ELIGIBILITY:
Inclusion Criteria:

* Consent form was signed by the individuals who accepted the study.

Exclusion Criteria:

* Individuals who smoke, who are pregnant, lactating and who are in the postmenopausal period, who take hormone therapy, who have followed any diet program for the last 3 months before the study, and who use vitamin/mineral supplementation were not included in the study.

Individuals who wanted to increase their physical activity level in addition to the applied diet were not included in the study.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 23 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-05-30 (Actual); Study Completion 2021-05-30 (Actual)

PRIMARY OUTCOMES:
Body weight in kilograms | 8 weeks
  Body weight measurement were taken using an Inbody 720 body analyzer.
The energy expenditure in kcal | 8 weeks
  Resting energy expenditure was measured at the beginning and end of the study using indirect calorimetry (COSMED, FitMatePro, Rome, Italy). Measurements were taken in the early morning hours after at least 8 hours of fasting.
Blood cholesterol level | 8 weeks
  The measurement was analyzed after at least 8 hours of fasting in the morning hours at the beginning and end of the study.
The quality of dietary intake | 8 weeks
  Diet quality was assessed with the Healthy Eating Index-2015 (HEI-2015).
Height in meters | 8 weeks
  The height of the individuals was measured with a stadiometer with a sensitivity of 0.1 cm.
waist circumference in meters | 8 weeks
  For waist circumference measurement, the midpoint between the lowest rib bone and the cristailiac was found, and the circumference measurement passing through this point was taken.
Blood Triglyceride level | 8 weeks
  The measurement was analyzed after at least 8 hours of fasting in the morning hours at the beginning and end of the study.
Blood fasting glucose level | 8 weeks
  The measurement was analyzed after at least 8 hours of fasting in the morning hours at the beginning and end of the study.
Blood insulin level | 8 weeks
  The measurement was analyzed after at least 8 hours of fasting in the morning hours at the beginning and end of the study.
Blood C-reactive protein level | 8 weeks
  The measurement was analyzed after at least 8 hours of fasting in the morning hours at the beginning and end of the study.
Blood leptin level | 8 weeks
  The measurement was analyzed after at least 8 hours of fasting in the morning hours at the beginning and end of the study.
Blood adiponectin level | 8 weeks
  The measurement was analyzed after at least 8 hours of fasting in the morning hours at the beginning and end of the study.
Blood total antioxidant status | 8 weeks
  The measurement was analyzed after at least 8 hours of fasting in the morning hours at the beginning and end of the study.
Blood total oxidant status | 8 weeks
  The measurement was analyzed after at least 8 hours of fasting in the morning hours at the beginning and end of the study.
Physical Activity Level (PAL) | 8 weeks
  Physical Activity Level (PAL) was determined by physical activity record.

CONTACTS AND LOCATIONS:
Overall Officials: ÖZGE MENGİ ÇELİK, Principal Investigator — University of Health science
Locations (1):
- Faculty of Health Science, Ankara, Turkey (Türkiye)